CLINICAL TRIAL: NCT05664763
Title: Understanding Effects of Cannabis Use and Abstinence on Neural Glutamate Homeostasis
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Stephen Baldassarri, Assistant Professor of Medicine, Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000033244; K23DA045957 (NIH)
Record Dates: First submitted 2022-12-14; First posted 2022-12-27 (Actual); Results first posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cannabis Use Disorder
Keywords: Cannabis; neuroimaging; marijuana; glutamate; tetrahydrocannabinol (THC)
MeSH Terms: conditions — Marijuana Abuse | interventions — 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabis use disorder (Experimental): CUD participants participants undergo neuroimaging, cognitive testing, and EEG at baseline and following cannabis abstinence at 4 weeks follow-up. Participants will receive motivational enhancement and contingency management during the 4-week abstinence period.
  Interventions: Drug: [18F]FPEB with PET; Behavioral: Cannabis abstinence
- Healthy control (Experimental): Healthy control participants undergo neuroimaging, cognitive testing, and EEG at baseline.
  Interventions: Drug: [18F]FPEB with PET

INTERVENTIONS:
Drug: [18F]FPEB with PET — radioactive tracer [18F]FPEB administered by bolus infusion over up to 2 hours with PET performed in the last 30 minutes of infusion with Positron emission tomography (PET) neuroimaging
Behavioral: Cannabis abstinence — Motivational enhancement and contingency management (CM) to promote and maintain cannabis abstinence after the baseline scan.
  Arms: Cannabis use disorder

SUMMARY:
This study will be the first in vivo human multimodal neuroimaging study exploring the relationship between mGluR5 availability (PET), neural oscillations (EEG), and cognitive function in people with CUD. The goal is to test the overall hypothesis that mGluR5 availability is higher in people with CUD compared with HC. In Aim 1, the investigators will determine differences in mGluR5 availability between people with CUD and HC in the fronto-limbic brain circuit. Aim 2 examines the associations between mGluR5 availability, CUD severity, neural oscillations, and cognitive function in CUD subjects. Aim 3 will determine how prolonged abstinence from chronic cannabis use affects mGluR5 availability, neural oscillations, and cognitive function in CUD subjects.

DETAILED DESCRIPTION:
Cannabis use and availability continue to rise significantly in the US. It is critical to expand our knowledge of the negative and positive effects of cannabis to "catch up" to the current reality of widespread and growing use. Cannabis and tetrahydrocannabinol (THC), its primary psychoactive chemical, have widespread effects on neural glutamate homeostasis, and specifically metabotropic glutamate receptor 5 (mGluR5). mGluR5 regulates transmission of glutamate and plays a critical role in neural plasticity (i.e., long-term potentiation; LTP), memory, learning, mood, and addiction. Specifically, it is thought that mGluR5 activation by glutamate initiates production of endocannabinoids (i.e., 2-AG) that bind retrograde to presynaptic cannabinoid receptor 1. This pathway inhibits further glutamate release and modulates synaptic plasticity diffusely in the brain. However, cannabis use disrupts this normal mechanism of glutamate homeostasis. While the relationship between cannabis use and glutamate regulation has been explored in preclinical models, it has not been well-characterized in humans, and particularly in people with cannabis use disorder (CUD).

The goal is to test the overall hypothesis that mGluR5 availability is higher in people with CUD compared with HC. This study will advance our understanding of cannabis effects on the neural glutamate system in humans and may lead to the development of novel therapeutics and biomarkers to treat people with CUD. Aim 1 will determine differences in mGluR5 availability between people with CUD and HC in the fronto-limbic brain circuit. Aim 2 examines the associations between mGluR5 availability, CUD severity, neural oscillations, and cognitive function in CUD subjects. Aim 3 will determine how prolonged abstinence from chronic cannabis use affects mGluR5 availability, neural oscillations, and cognitive function in CUD subjects.

ELIGIBILITY:
Inclusion Criteria:

HC and CUD Group:

* Voluntary, written, informed consent
* Physically healthy by medical history, physical, neurological, ECG and laboratory exams
* No personal or first-degree relative history of psychiatric disorders (outside of cannabis use for CUD group)
* Full scale and verbal IQs > 80 (Wechsler Adult Intelligence Scale, Fourth Edition; WAIS-IV).

CUD group:

* Cannabis use disorder as determined by DSM-5 structured interviews
* Urine toxicology evidence of cannabinoid use

HC group:

* lifetime cannabis exposure less than 20 times
* no cannabis use in the past 2 years by self-report
* a negative urine drug screen.

Exclusion Criteria:

* Other substance use disorder within 1 year, except for nicotine
* Another primary DSM-5 Axis I major psychiatric disorder (e.g., schizophrenia, bipolar disorder, major depression, etc.) per SCID-5
* Urine toxicology results positive for other drugs such as opiates / opiate metabolites (e.g., methadone, buprenorphine, etc.)
* A history of significant medical (cardiac, infectious, metabolic) or neurological illness (e.g., cerebrovascular disease, traumatic brain injury)
* A history of seizures/epilepsy
* Current use of psychotropic and/or potentially psychoactive prescription medications
* Medical contraindications to MRI imaging (e.g., ferromagnetic implants/foreign bodies, claustrophobia, etc.)
* Pregnancy or breastfeeding (women).
* Subjects will be excluded for major medical or neurological illness or laboratories consistent with these illnesses or suggesting contraindication to PET or MR imaging

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Baldassarri, M.D., Principal Investigator — Yale University
Locations (1):
- The Anlyan Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No healthy controls were enrolled.
Period: Overall Study
Arm/Group | Cannabis Use Disorder | Healthy Control
Started | 6 | 0
Only Attended One Visit | 3 | 0
Attended Both Visits | 3 | 0
Included in Analysis | 2 | 0
Completed | 3 | 0
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cannabis Use Disorder
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (6.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 1
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Metabotropic Glutamate Receptor 5 (mGluR5) Availability
Description: Participants will undergo a Positron Emission Tomography (PET) scan to visualized mGluR5 availability in the regions of interest (ROIs): orbitofrontal cortex (OFC), anterior cingulate, ventromedial prefrontal cortex (vmPFC), dorsolateral prefrontal cortex (dlPFC), hippocampus, and amygdala. Only done at baseline for HC group.
Time Frame: Baseline and Day 28
Measure: Mean (Standard Deviation); unit: ml/cm^3
Arm/Group | Cannabis Use Disorder
Number analyzed (Participants) | 2
ml/cm^3
  Amygdala | -2.218 (8.07)
  Anterior Cingulate | -4.03 (9.98)
  Dorsolateral Prefrontal Cortex | -3.94 (8.97)
  Hippocampus | -2.946 (7.21)
  Orbitofrontal Cortex | -5.2 (10.78)
  Ventromedial Prefrontal Cortex | -4.33 (9.97)

2. Secondary Outcome: Change in Neurocognitive Function Using CogState Cognitive Battery
Description: A battery of neuropsychological tests from the well-validated CogState Cognitive Battery are sensitive to detecting cognitive deficits in mood disorders, executive control and working memory. The entire battery takes approximately 30 minutes. Change in CUD group at baseline and day 28 compared to HC at baseline.
Time Frame: Baseline and Day 28
Population: Due to limitations in the availability of trained staff, data for the secondary outcomes were not collected. The project was scaled down to assess only the primary outcome, as reported above. All available data from this project have been reported. Data collection and analysis for this measure will not be conducted in the future.
Arm/Group | Cannabis Use Disorder
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Verbal Memory Measured Using Electroencephalography (EEG)
Description: Theta band power and coherence will be assessed. EEG data are collected in three separate conditions. In the passive listening condition, subjects will passively listen to a list of 15 words (presented one at a time) six times in a row. In the memory encoding condition, subjects will be administered a list of 15 words played one at a time, five times, and will be told to try and remember the list and to repeat as many words as possible after each list. Twenty minutes after the end of the encoding phase, subjects will be asked to repeat as many words as they can from the original list of words. In the computerized recognition condition, subjects will hear words from the (1) original memorized list, (2) the distractor list, and (3) novel words not heard that day. Subjects will respond with a three-choice button box to indicate from which list each word originated. Change in CUD group at baseline and day 28 compared to HC at baseline.
Time Frame: Baseline and Day 28
Population: as for outcome 2
Arm/Group | Cannabis Use Disorder
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Cannabis Use Disorder
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT05664763/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT05664763/ICF_001.pdf